CLINICAL TRIAL: NCT01744119
Title: Vascutek Anaconda™ Stent Graft System for Infra-Renal Abdominal Aortic Aneurysm Repair
Brief Title: Vascutek Anaconda™ Abdominal Aortic Aneurysm (AAA) Post-Market Surveillance Registry
Status: Terminated | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-PMS001
Record Dates: First submitted 2012-11-29; First posted 2012-12-06 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Abdominal Aortic Aneurysm
  Interventions: Device: Vascutek Anaconda™ Stent Graft System

INTERVENTIONS:
Device: Vascutek Anaconda™ Stent Graft System

SUMMARY:
The purpose of this observational Post-Market Surveillance Registry is to gather post-market data on the performance of the CE marked Vascutek Anaconda™ Stent Graft System for the repair of Abdominal Aortic Aneurysms (AAA). The Study population consists of patients suitable for endovascular repair of AAA. Patients will be followed at 1, 3, 6, 12, 18, 24, 36, 48 and 60 months post-implantation.

DETAILED DESCRIPTION:
Vascutek Limited, a world leader in the development of vascular grafts, has combined their latest technological developments in polyester textile technology with unique endovascular design features to produce Anaconda™, the world's next generation of AAA stent graft systems. Intuitive and of a modular design, Anaconda™ is the only repositionable device which also features exceptional flexibility. The modular design comprises bifurcate bodies, iliac legs and aortic cuffs. Nitinol, an alloy of nickel and titanium, has self-expanding properties and forms the top "ring-stent" of the bifurcate body section. The "ring stent" is composed of multiple turns of Nitinol wire that provides significantly increased "hoop-strength" enabling a conformable and secure haemostatic seal against the vessel wall to be achieved. Nitinol hooks located adjacent to the "ring stent" anchor the graft in position thus preventing graft migration. The iliac limbs are fully supported with Nitinol and the bifurcate bodies feature a distal contra-lateral lumen Nitinol support, which in conjunction with a unique intrinsic magnet guidewire system facilitates cannulation of the bifurcate section.

The system is available in a wide range of sizes thus making it a flexible and adaptable stent graft system with the potential to repair diverse patient anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is implanted with Anaconda™ Stent Graft System

Exclusion Criteria:

* Ruptured or symptomatic aneurysm
* Juxta or Suprarenal extension of aneurysm
* Clinically serious concomitant medical disease or infection
* Need to sacrifice both Internal Iliac Arteries due to aneurysmal dilatation
* Connective Tissue Disease (Marfan's Syndrome)
* ASA Rating of Grade IV or V
* Known allergy to Nitinol, Polyester or contrast medium
* Excessive tortuosity of access vessels (femoral or iliac arteries)
* Patients with aneurysm neck lengths of less than 15mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a CE-Marked Vascutek Anaconda™ Stent Graft System for Infra-Renal Abdominal Aortic Aneurysm Repair
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2005-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of graft performance | 60 months
  Data will be collected and analysed on system insertion and difficulty during deployment. Efficiency of the magnet system including magnet selection, ease of use and removal of magnet guidewire will also be evaluated.
Graft patency | 60 months
  Data will be collected and analysed on endoleak exclusion and graft migration rates
Exclusion of aneurysm | 60 months

CONTACTS AND LOCATIONS:
Locations (21):
- Australia (7):
  - Dalcross Private Hospital, Killara, New South Wales
  - Newcastle Private Medical Suites, Newcastle, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Austin Hospital, Heidelberg, Victoria
  - Geelong Regional Vascular Service, Geelong
  - Royal Perth Hospital, Perth
  - Hollywood, Royal Perth, Perth
- Clinique Guillaume De Varye, Saint-Doulchard, France
- Germany (3):
  - DRK Kliniken Mark Brandenburg, Berlin
  - Dresden-Friedrichstadt, Dresden
  - Klinikum Grosshadern, Munich
- Italy (4):
  - San Orsola - Bologna University, Bologna
  - University federico II, Naples
  - Guglielmo da Saliceto, Piacenza
  - Casa di Cura Nuova Itor, Roma
- New Zealand (2):
  - Christchurch Hospital, CDHB, Christchurch
  - Waikato Hospital, Hamilton
- Hospital Universitario Madrid Monteprincipe, Madrid, Spain
- United Kingdom (3):
  - Royal Derby Hospital, Derby
  - Gartnavel General Hospital, Glasgow
  - Wishaw General Hospital, Wishaw